CLINICAL TRIAL: NCT03208738
Title: Pilot Evaluation of the VetChange Mobile App for Veterans With PTSD Who Engage in Problem Drinking
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Eric Kuhn (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Eric Kuhn, Clinical Psychologist, VA Palo Alto Health Care System
Organization: VA Palo Alto Health Care System (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-38085
Record Dates: First submitted 2017-06-30; First posted 2017-07-05 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Alcohol Abuse; Post-Traumatic Stress Disorder
MeSH Terms: conditions — Alcoholism; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Masking Description: NA: All study measures are self-report.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Assessment only (No Intervention)
- VetChange mobile app (Experimental)
  Interventions: Behavioral: VetChange
- AFT + VetChange mobile app + supportive accountability tool (Experimental)
  Interventions: Behavioral: VetChange; Behavioral: web-based drinking assessment and feedback tool (AFT)

INTERVENTIONS:
Behavioral: VetChange — VetChange is a self-management mobile application designed to to concurrently reduce both alcohol misuse and PTSD symptoms.
  Arms: AFT + VetChange mobile app + supportive accountability tool; VetChange mobile app
Behavioral: web-based drinking assessment and feedback tool (AFT) — Program will administer a comprehensive assessment of drinking and consequences of drinking, and will provide normative feedback and highlight negative consequences of drinking.
  Arms: AFT + VetChange mobile app + supportive accountability tool

SUMMARY:
Concept: Alcohol misuse is common among Veterans with PTSD. It has been proposed that this high comorbidity is the result of "self-medication," with alcohol being used to alleviate common PTSD symptoms (e.g., hyperarousal, sleep problems). Given this high prevalence and functional relationship, researchers at the BSD of the NCPTSD developed the VetChange self-management website to concurrently address these conditions. In a large scale RCT, VetChange has shown efficacy to reduce both alcohol misuse and PTSD symptoms. Unfortunately, the recently launched publicly available VetChange website (Vetchange.org) has been plagued by a high rate of visitors not completing the mandatory registration process, which is required for repeated use. Based on the promising findings of the VetChange research, the D&T Division partnered with the BSD Division to develop the VetChange mobile app, which is set to be released to the public very soon. However, unlike the VetChange website, the app has not yet been evaluated and has the advantage of allowing users to easily obtain it without having to register and repeatedly log on through an Internet connection.

This research partnership between the D&T and BSD Divisions will extend and enhance an ongoing successful cross-center collaboration in a high priority topic for the larger Center. The purpose of this proposal is to conduct a pilot evaluation of the VetChange mobile app in order to test its feasibility, acceptability, and potential efficacy to reduce alcohol consumption, PTSD severity, and improve psychosocial functioning among Veterans with PTSD who exhibit signs of problem drinking. In this study, 280 Veterans with problem drinking and clinically significant PTSD symptoms will be recruited using social media and randomized in equal numbers to receive one of four conditions: 1) Assessment only, 2) VetChange mobile app only, 3) AFT plus the VetChange mobile app supplemented with a package of supportive accountability tools (VetChange+). In addition to receiving the mobile app, VetChange+ participants will receive SMS reminders to log drinking behavior using the mobile app. The investigators will track objective use of the VetChange mobile app to assess feasibility, and this usage data will also be used in real-time to tailor the content of text messages provided to participants in the VetChange+ condition. Participants will complete measures of alcohol use, functional well-being, and PTSD symptoms at baseline and again after 8 weeks (posttreatment). At post-treatment, participants in the VetChange app arms of the study will also be asked to report their level of satisfaction with the app and to complete a brief qualitative evaluation of their experience using the VetChange mobile app.

Results of this pilot study will be used to characterize the feasibility, acceptability, and potential efficacy of a mobile app-based self-management intervention to reduce problem drinking behavior in Veterans with PTSD, will inform optimization of the intervention, and will serve as the foundation for subsequent proposals for extramural funding.

ELIGIBILITY:
Inclusion Criteria:

1. self-reported status as OEF or OIF veteran,
2. age between 18 and 65 years,
3. moderate levels of nondependent problem drinking as determined by score on the Alcohol Use Disorders Identification Test (AUDIT; Babor, de la Fuente, Saunders, & Grant, 1992; Bradley et al., 2003) between 8 and 25 for men and 5 and 25 for women,
4. drinking above guidelines for safer drinking during the 30 days prior to screening based on the Quick Drink Screen (L. C. Sobell et al., 2003; no more than 4 drinks per occasion or 14 drinks per week for men and no more than three drinks per occasion or seven drinks per week for women; Dawson, Grant, & Li, 2005; U.S. Department of Health and Human Services & U.S. Department of Agriculture, 2010), and
5. willing to provide an e-mail address for reminders and incentives.

Exclusion Criteria:

(a) high alcohol problem severity

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2017-07 (Estimated); Primary Completion 2018-06 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Quick Drink Screen (QDS; Sobell et al., 2003) | 8 weeks
  4-item self-report measure of alcohol consumption focused on quantity and frequency of drinking in the last 30 days
PTSD Checklist-5 (PCL-5; Weathers et al., 2010) | 8 weeks
  20-item self-report measure of PTSD symptoms

SECONDARY OUTCOMES:
The Short Inventory of Problems (SIP; Miller, Tonigan, & Longabaugh, 1995) | 8 weeks
  15-item, self-report of alcohol-related problems